CLINICAL TRIAL: NCT05744063
Title: An Open Label, Single Arm, Multi-Centre, Post-authorization Study to Describe the Safety and Efficacy of Emapalumab for the Treatment of Primary Hemophagocytic Lymphohistiocytosis in Treatment Experienced Chinese Patients
Brief Title: A Post-authorization Study to Describe the Safety and Efficacy of Emapalumab for the Treatment of pHLH in Treatment Experienced Chinese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.emapalumab-104
Record Dates: First submitted 2023-02-13; First posted 2023-02-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Primary Hemophagocytic Lymphohistiocytosis
Keywords: pHLH
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Emapalumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, multi-centre study to collect safety and efficacy data on emapalumab in treatment experienced male and female patients diagnosed with pHLH. The study will be performed in China.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- emapalumab (Experimental): emapalumab solution for infusion twice weekly at a starting dose of 1 mg/kg
  Interventions: Drug: Emapalumab-Lzsg 5 MG/ML [Gamifant]

INTERVENTIONS:
Drug: Emapalumab-Lzsg 5 MG/ML [Gamifant] — iv
  Other Names: Gamifant

SUMMARY:
The goal of this post-authorization study is to describe safety and efficacy of emapalumab in treatment experienced Chinese patients with pHLH.

DETAILED DESCRIPTION:
This is an open-label, multi center, single arm, post-authorization study aiming to describe safety and efficacy of emapalumab in treatment experienced Chinese patients with confirmed or suspected primary hemophagocytic lymphohistiocytosis (pHLH). The main objectives of the study are to collect safety and efficacy data on emapalumab in treatment experienced Chinese pHLH patients

ELIGIBILITY:
Inclusion Criteria:

1. Male and female HLH patients of any age.
2. Patients diagnosed with confirmed or suspected pHLH, based on; a molecular diagnosis or familial history consistent with pHLH or fulfilment of HLH-2004 diagnostic criteria, i.e., five out of eight of the criteria below:

   * Fever
   * Splenomegaly
   * Cytopenias affecting 2 of 3 lineages in the peripheral blood (hemoglobin <90 g/L; platelets <100 x 109/L; neutrophils <1 x 109/L)
   * Hypertriglyceridemia (fasting triglycerides ≥3 mmol/L or ≥265 mg/dL) and/or hypofibrinogenemia (≤1.5 g/L)
   * Hemophagocytosis in bone marrow, spleen, or lymph nodes, with no evidence of malignancy.
   * Low or absent NK-cell activity
   * Ferritin ≥500 μg/L
   * Soluble CD25 (sCD25; i.e., soluble IL-2 receptor) ≥2400 U/mL
3. Presence of active HLH disease as assessed by the investigator.
4. Patients must fulfil one of the following criteria as assessed by the investigator:

   * Having not responded to previous conventional treatment of HLH
   * Having not achieved a satisfactory response to previous conventional treatment of HLH or worsened
   * Having reactivated HLH
   * Showing intolerance to previous conventional treatment of HLH At the time of enrollment, eligible patients might still be receiving treatment (induction or maintenance) or might have already discontinued it.
5. Expectation of survival beyond 1 week as judged by the investigator.
6. Patient has expectation of proceeding to HSCT
7. Informed consent signed by the patient (as required by local law), or by the patient's legally authorized representative(s) with the assent of patients who are legally capable of providing it, as applicable.
8. Willing to use highly effective methods of contraception from study drug initiation to 6 months after the last dose of study drug, if female and of childbearing potential.

Exclusion Criteria:

1. Diagnosis of secondary HLH consequent to a proven rheumatic, metabolic or neoplastic disease.
2. Active mycobacteria, Histoplasma capsulatum, Salmonella, or Leishmania infections.
3. Evidence of latent tuberculosis.
4. Presence of malignancy.
5. Existence of any severe co-morbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for the treatment
6. History of hypersensitivity or allergy to any component of the study regimen (e.g., polysorbate).
7. Receipt of a Bacillus Calmette-Guérin (BCG) vaccine within 12 weeks prior to Screening.
8. Receipt of a live or attenuated live (other than BCG) vaccine within 4 weeks prior to Screening.
9. Pregnant or lactating female patients.
10. Enrollment in another concurrent clinical interventional study, or intake of an IMP, within three months prior to inclusion in this study
11. Any condition or circumstance that in the opinion of the Investigator may make the patient unlikely to complete the study or comply with study procedures or requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Permanent discontinuation of study drug due to emapalumab-related adverse event | until conditioning for hematopoietic stem cell transplant (HSCT), likely within 6 months from first dose
  as judged by Investigator

SECONDARY OUTCOMES:
Overall response | end of treatment or week 8 (whichever occurs earlier)
  measured as complete response, partial response, or HLH improvement
Time to first overall response | end of treatment, likely within 6 months from first dose
  from first dose of study drug to first response
Cumulative duration of response | end of treatment, likely within 6 months from first dose
  total time in response
Ability to reduce glucocorticoids by 50% or more | end of treatment, likely within 6 months from first dose
  reduction from baseline dose during emapalumab treatment
Investigator assessed response | end of treatment or week 8 (whichever occurs earlier)
  Investigator's assessment of how patient responds to treatment and rated as complete response, partial response, or no response
Survival | end of study
  To start of HSCT conditioning and after time from HSCT to death

CONTACTS AND LOCATIONS:
Overall Officials: Rui Zhang, MD, Prof, Principal Investigator — Beijing Children's Hospital
Locations (7):
- China (7):
  - Swedish Orphan Biovitrum Research site, Shanghai, Fudan
  - Swedish Orphan Biovitrum Research site, Beijing, Xicheng
  - Swedish Orphan Biovitrum Research site, Beijing
  - Swedish Orphan Biovitrum Research site, Chongqing
  - Swedish Orphan Biovitrum Research site, Guangzhou
  - Swedish Orphan Biovitrum Research site, Nanjing
  - Swedish Orphan Biovitrum Research site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No